CLINICAL TRIAL: NCT01310140
Title: Comparative Risks for Insulin Resistance and Metabolic Syndrome (MS) Among Hospitalized Patients With Major Depressive Disorder With (MDpsy) or Without (MDD) Psychotic Features
Brief Title: Risks for Insulin Resistance and Metabolic Syndrome Between Major Depressive Disorder (MDD) or MDD With Psychotic Features
Status: Terminated | Type: Observational
Why Stopped: PI left Massachusetts General Hospital Inpatient service
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, John D. Matthews, Principal Investigator, Assistant Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2009-P-002723
Record Dates: First submitted 2011-02-15; First posted 2011-03-08 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Major Depressive Disorder; Major Depressive Disorder w/ Psychotic Features; Metabolic Syndrome
Keywords: Metabolic Syndrome; Insulin Resistance; Massachusetts General Hospital; Major Depressive Disorder; Major Depressive Disorder with Psychotic Features; Cortisol; Dexamethasone Suppression Test
MeSH Terms: conditions — Depressive Disorder, Major; Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Major Depressive Disorder
- Major Depressive Disorder with Psychotic Features

SUMMARY:
Studies have shown that people with certain disorders have an increased risk of developing a condition called Metabolic Syndrome (MS). In this study, the investigators want to learn more about MS among people staying in the hospital for treatment of Major Depressive Disorder (MDD) and also Major Depressive Disorder with Psychotic Features (MDpsy). The investigators also want to learn more about a stress hormone called cortisol that is made in the body. Those who take part in this study will answer some questionnaires, be given some psychiatric interviews, and have some blood taken along with a urine sample.

The investigators believe that patients in the hospital with MDpsy will have higher baseline rates of MS factors, cortisol levels, dexamethasone non-suppression, and insulin resistance, compared with MDD alone.

DETAILED DESCRIPTION:
Metabolic syndrome (MS) is a combination of medical problems that can increase the risk of heart disease and diabetes in some people. People with MS can have some or all of the following:

* High blood glucose
* High blood pressure
* Abdominal obesity
* Low levels of high-density lipoprotein (HDL) cholesterol
* High levels of triglycerides

Some studies have shown that people with certain disorders have a greater risk for developing MS. This may be because of a combination of factors, including but not limited to the type of medications used, age, and whether or not someone smokes. This study will also aim to learn more about a naturally-occurring stress hormone called cortisol that is made in the body.

In order to measure these factors, the following things will occur:

* administer a number of questionnaires
* gather information from medical history
* gather information about current psychiatric mood
* draw blood and collect a urine sample

To study the amount of cortisol in the body, a dexamethasone suppression test (DST) will be given. This test involves taking a single 1mg pill of dexamethasone, a steroid, and numerous blood draws. Like any drug, it has some risks, however it is unlikely any side effects will occur because of the low dose administered.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* DSM-IV TR diagnosis of Major Depressive Disorder with (MDpsy) or without (MDD) Psychotic Features
* Age between 18 and 85, inclusive
* Pre-existing Hyperlipidemia, Hypertension, and Diabetes must be stable with laboratory and clinical results within acceptable range; with or without medication for three months prior to admission

Exclusion Criteria:

* DSM-IV TR diagnosis of: schizophrenia, schizoaffective disorder, delusional disorder, bipolar disorder, organic mental disorder, substance use dependence including alcohol, that has been active within the past 6 months, acute bereavement, and psychotic disorder not elsewhere classified
* Subjects that meet criteria for substance or alcohol dependence more recently than three months prior to entering the study
* Subjects that meet criteria for substance or alcohol abuse more recently than four weeks prior to entering the study
* Pregnancy
* Unstable or inadequately treated pre-existing hyperlipidemia, hypertension, and diabetes
* Subjects who are involuntarily committed.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects are people who are inpatient in the medical-psychiatric unit at Massachusetts General Hospital. Included subjects have working diagnosis of major depressive disorder (MDD) or major depressive disorder with psychotic features (MDpsy).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The primary measure is any change in fasting insulin from admission to discharge while subjects are inpatient. | Measure fasting insulin at two timepoints; to determine change from baseline (admission) and discharge
  To preserve statistical power, we will measure insulin as a continuous variable rather than dichotomizing participants into insulin sensitive vs insulin resistant.

SECONDARY OUTCOMES:
The first secondary measure is a fasting lipid panel, including fasting total cholesterol, fasting LDL, fasting HDL, and fasting triglycerides; we want to measure a change in data from admission to discharge | Two separate timepoints during inpatient hospitalization; first within 5 days of admission, and second within 72 hours of scheduled discharge
Fasting glucose will be a separate secondary outcome measure; we want to measure a change in data from admission to discharge | Two separate timepoints during inpatient hospitalization; first within 5 days of admission, and second within 72 hours of scheduled discharge
Waist Circumference; we want to measure a change in data from admission to discharge | Two separate timepoints during inpatient hospitalization; first within 5 days of admission, and second within 72 hours of scheduled discharge
  Waist circumference will be measured once at admission and once at discharge to determine if any changes have occurred throughout time of inpatient hospitalization
Urine microalbumin; we want to measure a change in data from admission to discharge | Two separate timepoints during inpatient hospitalization; first within 5 days of admission, and second within 72 hours of scheduled discharge
C-reactive Protein; we want to measure a change in data from admission to discharge | Two separate timepoints during inpatient hospitalization; first within 5 days of admission, and second within 72 hours of scheduled discharge
Homocysteine; we want to measure a change in data from admission to discharge | Two separate timepoints during inpatient hospitalization; first within 5 days of admission, and second within 72 hours of scheduled discharge
Blood pressure (supine & standing as available) | We will be measuring this continuously throughout inpatient hospitalization, beginning at time of admission
Cortisol; we want to measure a change in data from admission to discharge | Two separate timepoints during inpatient hospitalization; first within 5 days of admission, and second within 72 hours of scheduled discharge
  Cortisol levels will be measured before and after a dexamethasone suppression test is administered at admission and discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States